CLINICAL TRIAL: NCT00810745
Title: What Benefit With a New Stapler Device in the Surgical Treatment of Obstructed Defecation? Two-Year Outcomes From a Randomized Controlled Trial
Brief Title: What Benefit With a New Stapler Device in the Surgical Treatment of Obstructed Defecation?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: first department of general surgery, university of milan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: starr
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Rectal Prolapse
Keywords: ODS; stapled transanal rectal resection
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- rectal resection (Experimental)
  Interventions: Procedure: starr

INTERVENTIONS:
Procedure: starr — stapled transanal rectal resection

SUMMARY:
This randomized study was designed to compare the 2 year clinical and functional results with the STARR procedure using a new curved cutter stapler or the same operation done with 2 traditional circular staplers.

DETAILED DESCRIPTION:
From January to November 2006, 80 women were selected, with clinical examination, constipation score, colonoscopy, anorectal manometry, and perineography and randomly assigned to 2 groups: 40 patients underwent stapled transanal rectal resection with two staplers PPH-01 (Ethicon Endosurgery Inc, Pomezia, Italy) (STARR group) and 40 had the same operation with new, curved multi-fire stapler Contour R Transtar TM (TRANSTAR group). Patients were followed up with clinical examination, constipation score, and perineography.

ELIGIBILITY:
Inclusion Criteria:

* Rectal prolapse
* Rectocele
* ODS score > 15
* Continence score < 3
* Resting pressure > 40 mm/Hg

Exclusion Criteria:

* Previous anorectal surgery
* Ods score < 15
* Continence score > 3
* Resting pressure < 40
* Concomitant pelvic floor diseases
* Psychiatric diseases
* Absolute contraindications to surgery

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-01; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
incidence of recurrences | 2 years

SECONDARY OUTCOMES:
outcomes on symptoms and defecography | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: paolo boccasanta, md, Principal Investigator — 1 department of general surgery
Locations (2):
- Italy (2):
  - First department of general surgery university of milan, Milan
  - First Department of General Surgery, Milan